CLINICAL TRIAL: NCT07099664
Title: Use of the Aortic Time-velocity Integral (VTI) Via Suprasternal Ultrasound to Search Preload Dependence in Paediatric Surgery : Kid's Fluid Management (FM)
Brief Title: Use of the Aortic Time-velocity Integral Via Suprasternal Ultrasound to Search Preload Dependence in Paediatric Surgery : Kid's Fluid Management (FM)
Acronym: Kid's FM
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_0708; 2024-A01473-44 (Other: ID-RCB Number)
Record Dates: First submitted 2025-06-30; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Hemodynamic
Keywords: Suprasternal doppler; paediatric anaesthesia; hemodynamic; fluid management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Measurement of VTI variation and cardiac output after general anaesthesia.: Measurement of VTI variation and cardiac output after general anaesthesia. Patients responding to volume expansion (more than 10% increase of cardiac output measured by transthoracic ultrasound after a 10ml/kg perfusion of cristalloids)
  Interventions: Diagnostic Test: Measurement of aortic Vmax and VTI with suprasternal doppler.

INTERVENTIONS:
Diagnostic Test: Measurement of aortic Vmax and VTI with suprasternal doppler. — Measurement of aortic Vmax and VTI with suprasternal doppler. Measurement of VTI variation and cardiac output after general anaesthesia. After preoperative fasting compensation, measurement of cardiac output (CO). Search of a difference in the suprasternale VTI variability between the patients who have increased their CO after fasting compensation and the patient who haven't.

SUMMARY:
After major surgery, fluid overload is associated with an increase of morbidity and mortality.

Fluid administration should therefore be given wisely. However, there is a paucity of monitor to predict preload dependence in paediatric anaesthesia.

The aim of this study is to determine if VTI variation, measured through the suprasternal window, with a cardiac doppler probe, can predict preload dependence.

Indeed, cardiac probe are present in most operating room and suprasternal window is reachable in most surgical case, which should allow VTI monitoring for the vast majority of our patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient under 18 admitted to paediatric operating room for a surgical intervention, an endoscopy, an interventional radiology procedure or an imagery and needing a general anaesthesia.

Exclusion Criteria:

* Condition preventing a suprasternal ultrasound (tracheostomy, spinal immobilization, suprasternal bandage)
* Pathology disturbing respiratory variation of left ventricular stroke volume (PAH, constrictive pericarditis, pericardial effusion, right ventricular dysfunction, complex congenital heart disease, aortic coarctation, patent ductus arteriosus
* Every medical condition where Berry's rule of fasting compensation could be unsafe (anuric kidney failure, oedema, heart failure with reduce left ventricular ejection fraction, patient under vasoactive drugs
* Opposition to the participation in the study
* Pregnant women
* Patient with no security coverage
* Inability to determine baseline cardiac output

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patient under 18 admitted to paediatric operating room for a surgical intervention, an endoscopy, an interventional radiology procedure or an imagery and needing a general anaesthesia
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Aortic VTI variation (%) measured by suprasternal doppler in percent of mean aortic VTI. | During preoperative, after induction and fasting compensation, before incision.

SECONDARY OUTCOMES:
Proportion of patient (%) in whom we can use suprasternal aortic measurements. | During preoperative period, after induction and fasting compensation, before incision.
Optimal threshold of aortic VTI variation (%) measured by suprasternal doppler to determine wether the patient is preload dependant or independent as defined above. | During preoperative period, after induction and fasting compensation, before incision.
  Optimal threshold of aortic VTI variation (%) measured by suprasternal doppler to determine wether the patient is preload dependant or independent as defined above (more than 10% increase of cardiac output measured by transthoracic ultrasound after a 10mL/kg perfusion of cristalloids OR not).
Correlation between : - fasting duration in hours, determined by patient or parent interrogation. - preload dependence as defined above. More than one outcome measure appears to be described. | During preoperative period, after induction and fasting compensation, before incision.
  Correlation between :
  * fasting duration in hours, determined by patient or parent interrogation.
  * preload dependence as defined above (increase of 10% or more of stroke volume measured by transthoracic ultrasound after a 10mL/kg perfusion of cristalloids).
  More than one outcome measure appears to be described.

IPD SHARING:
Plan to Share IPD: No